CLINICAL TRIAL: NCT02659436
Title: Imagery-based CBT for Social Anxiety Disorder: Piloting a Treatment Augmentation Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Karen Rowa, Associate Professor and Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0986
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Social Anxiety Disorder
Keywords: Cognitive Behavioural Therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verbal-linguistic CBT (Active Comparator): Participants will receive 4 sessions of verbal cognitive restructuring and exposure therapy delivered in an individual therapy format.
  Interventions: Other: Verbal-linguistic CBT
- Imagery-based CBT (Experimental): Participants will receive 4 sessions of imagery-based cognitive work and behavioural experiments delivered in an individual therapy format.
  Interventions: Other: Imagery-based CBT

INTERVENTIONS:
Other: Verbal-linguistic CBT — Participants will receive 4 sessions of individual therapy focused on traditional cognitive restructuring and exposure therapy.
  Arms: Verbal-linguistic CBT
Other: Imagery-based CBT — Participants will receive 4 sessions of individual therapy focused on imagery-based cognitive work and behavioural experiments.
  Arms: Imagery-based CBT

SUMMARY:
The purpose of this pilot study is to explore whether there is a differential impact of verbal versus imagery-based cognitive behavioural therapy (CBT) as a treatment augmentation strategy for individuals with social anxiety disorder (SAD). Clients who have not demonstrated clinically significant change following group CBT for SAD will receive four additional sessions of either verbal-based CBT or imagery-based CBT. We hypothesize that that individuals who receive imagery-based CBT will experience even stronger improvements and be more satisfied with their treatment than individuals who received traditional verbal-linguistic CBT.

DETAILED DESCRIPTION:
Social Anxiety Disorder (SAD) is a debilitating disorder, marked by significant functional impairment and high personal distress for those who suffer. Psychological treatment for SAD has traditionally been verbal-linguistic cognitive behavioural therapy (CBT). However, a significant number of individuals who complete CBT for SAD do not achieve full response and continue to struggle with significant residual symptoms. One innovation that has received attention recently in the literature is using imagery-based CBT as a way to augment treatment outcome in SAD. Results from a pilot and benchmarking study suggest that participants who received imagery-based CBT were more likely to complete treatment than those who received traditional CBT and treatment outcome was strong for both groups, but stronger in the imagery-based CBT group.

However, before re-training hundreds of practitioners in using a completely novel treatment approach, it is important to see if a brief augmentation of traditional CBT programs is effective in producing further change for individuals with residual symptoms after group CBT. It is possible that individuals just require a few more sessions of the same verbal-linguistic CBT to consolidate treatment gains or work on lingering triggers of anxiety. It is also possible that more of the same is not as valuable as offering therapy using a different modality, such as imagery. Therefore, we propose to evaluate a brief imagery-based augmentation of traditional group CBT to explore its effects on further symptom reduction.

ELIGIBILITY:
Inclusion Criteria:

* Completed eight out of twelve sessions of standard verbal-linguistic group cognitive behavioural therapy for social anxiety disorder
* Presented with a Social Phobia Inventory (SPIN) score of greater than 19 post-treatment
* Interested in further treatment

Exclusion Criteria:

* Has another mental health concern of greater importance than social anxiety disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Social Phobia Inventory | This will be administered at the end of the 4 session protocol which will take place approximately 4 -6 weeks after entry into the study.
  Measures social anxiety symptoms

SECONDARY OUTCOMES:
Vividness of Visual Imagery Questionnaire | This will be administered at the end of the 4 session protocol which will take place approximately 4 -6 weeks after entry into the study.
  Measures the ability to visualize several visual images
Homework Adherence Scale | This will be administered at the end of the 4 session protocol which will take place approximately 4 -6 weeks after entry into the study.
  Measures the quality of homework completion
Treatment Satisfaction Scale | This will be administered at the end of the 4 session protocol which will take place approximately 4 -6 weeks after entry into the study.
  Measures the participant's satisfaction with their treatment
Brief Fear of Negative Evaluation Scale | This will be administered at the end of the 4 session protocol which will take place approximately 4 -6 weeks after entry into the study.
  Measures fears about being negatively evaluated by others
Illness Intrusiveness Rating Scale | This will be administered at the end of the 4 session protocol which will take place approximately 4 -6 weeks after entry into the study.
  Measures how much anxiety interferes with functioning

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rowa, Ph. D, Principal Investigator — St. Joseph's Healthcare Hamilton

REFERENCES:
- [Background] American Psychiatric Association (2013). Diagnostic and statistical manual of mental disorders (5th edition). Washington, DC: APA.
- [Background] Antony MM, Roth D, Swinson RP, Huta V, Devins GM. Illness intrusiveness in individuals with panic disorder, obsessive-compulsive disorder, or social phobia. J Nerv Ment Dis. 1998 May;186(5):311-5. doi: 10.1097/00005053-199805000-00008. PMID 9612449
- [Background] Bieling, P.J., Rowa, K., Antony, M.M., Summerfeldt, L.J., & Swinson, R.P. (2001). Factor structure of the Illness Intrusiveness Ratings Scale in patients diagnosed with anxiety disorders. Journal of Psychopathology and Behavioral Assessment, 23, 223-230. doi: 10.1023/A:1012723318964
- [Background] Carleton RN, Collimore KC, Asmundson GJ. Social anxiety and fear of negative evaluation: construct validity of the BFNE-II. J Anxiety Disord. 2007;21(1):131-41. doi: 10.1016/j.janxdis.2006.03.010. Epub 2006 May 3. PMID 16675196
- [Background] Devins GM. Illness intrusiveness and the psychosocial impact of lifestyle disruptions in chronic life-threatening disease. Adv Ren Replace Ther. 1994 Oct;1(3):251-63. doi: 10.1016/s1073-4449(12)80007-0. PMID 7614328
- [Background] Devins GM, Dion R, Pelletier LG, Shapiro CM, Abbey S, Raiz LR, Binik YM, McGowan P, Kutner NG, Beanlands H, Edworthy SM. Structure of lifestyle disruptions in chronic disease: a confirmatory factor analysis of the Illness Intrusiveness Ratings Scale. Med Care. 2001 Oct;39(10):1097-104. doi: 10.1097/00005650-200110000-00007. PMID 11567172
- [Background] Hackmann A, Clark DM, McManus F. Recurrent images and early memories in social phobia. Behav Res Ther. 2000 Jun;38(6):601-10. doi: 10.1016/s0005-7967(99)00161-8. PMID 10846808
- [Background] Hirsch CR, Clark DM, Mathews A, Williams R. Self-images play a causal role in social phobia. Behav Res Ther. 2003 Aug;41(8):909-21. doi: 10.1016/s0005-7967(02)00103-1. PMID 12880646
- [Background] Holmes EA, Lang TJ, Shah DM. Developing interpretation bias modification as a "cognitive vaccine" for depressed mood: imagining positive events makes you feel better than thinking about them verbally. J Abnorm Psychol. 2009 Feb;118(1):76-88. doi: 10.1037/a0012590. PMID 19222316
- [Background] Leary, M. R. (1983). A brief version of the Fear of Negative Evaluation Scale. Personality and Social Psychology Bulletin, 9, 371-376. doi: 10.1177/0146167283093007
- [Background] McEvoy PM, Saulsman LM. Imagery-enhanced cognitive behavioural group therapy for social anxiety disorder: a pilot study. Behav Res Ther. 2014 Apr;55:1-6. doi: 10.1016/j.brat.2014.01.006. Epub 2014 Feb 7. PMID 24561919
- [Background] McEvoy PM, Erceg-Hurn DM, Saulsman LM, Thibodeau MA. Imagery enhancements increase the effectiveness of cognitive behavioural group therapy for social anxiety disorder: a benchmarking study. Behav Res Ther. 2015 Feb;65:42-51. doi: 10.1016/j.brat.2014.12.011. Epub 2014 Dec 27. PMID 25569339
- [Background] Moscovitch DA, Gavric DL, Merrifield C, Bielak T, Moscovitch M. Retrieval properties of negative vs. positive mental images and autobiographical memories in social anxiety: outcomes with a new measure. Behav Res Ther. 2011 Aug;49(8):505-17. doi: 10.1016/j.brat.2011.05.009. Epub 2011 May 26. PMID 21683343